CLINICAL TRIAL: NCT03384511
Title: Whether 18F-ALF-NOTA-PRGD2 PET/CT Scan Can Predict the Efficacy and Adverse Events of Apatinib in Patients With Malignancies.
Brief Title: The Use of 18F-ALF-NOTA-PRGD2 PET/CT Scan to Predict the Efficacy and Adverse Events of Apatinib in Malignancies.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, ShuanghuYuan, M.D., Ph.D., Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRTOG1701
Record Dates: First submitted 2017-09-01; First posted 2017-12-27 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Malignancies; Stomach Cancer; Non-small Cell Lung Cancer; Esophageal Cancer; Breast Cancer; Ovary Cancer; Cervical Cancer
Keywords: RGD PET-CT; Apatinib
MeSH Terms: conditions — Neoplasms; Stomach Neoplasms; Carcinoma, Non-Small-Cell Lung; Esophageal Neoplasms; Breast Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms | interventions — apatinib

STUDY DESIGN:
Intervention Model Description: Apatinib at oral dose of 250 mg twice daily (500 mg/day) for a minimum of 30 days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Apatinib & RGD PET/CT (Experimental): All of the patients will receive apatinib at oral dose of 250 mg twice daily (500 mg/day) at least 30 days.One treatment cycle is defined as 4 weeks.18F-ALF-NOTA-PRGD2 PET/CT scan will be performed berore and after one cycle of therapy. Treatment interruptions or dose reductions to 250 mg/day will be allowed for the management of adverse events. The maximum allowable period of treatment interruption is 1 week during each treatment cycle, and the dose should be re-escalated to 500 mg/day after adverse events mitigation. Treatment will not stop until disease progression, intolerable toxicity, or patients' request for withdrawal from the study.
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Patients will accept apatinib therapy and undergo baseline 18F-ALF-NOTA-PRGD2 PET/CT scans of the whole body after having met all eligibility criterias.
  Other Names: YN968D1

SUMMARY:
This is an open-label, single arm study to explore whether 18F-ALF-NOTA-PRGD2 PET/CT scan can predict the efficacy and adverse events of apatinib in patients with malignancies.

Integrin αvβ3 has been shown to play an important role in angiogenesis and up-regulated obviously in various types of tumor cells and activated endothelial cells. The arginine-glycine-aspartic acid (RGD) tripeptide sequence can bind to integrin αvβ3 with high affinity and specificity. The 18F-ALF-NOTA-PRGD2 will highly combine with αvβ3, and thus will monitor the antiangiogenic status.In the current study, investigators propose to evaluate the feasibility of 18F-RGD PET/CT in monitoring efficacy and adverse events of apatinib in malignancies.

DETAILED DESCRIPTION:
This is an open-label, single arm study to explore whether 18F-ALF-NOTA-PRGD2 positron emission tomography/computed tomography (18F-RGD PET/CT) scan can predict the efficacy and adverse events of apatinib in patients with malignancies.

Angiogenesis, the formation of new blood vessels, is the process of generating neovascularization from preexisting vessels. It can promote tumor growth and metastasis by providing nutrients and oxygen. Integrin αvβ3 has been shown to play an important role in angiogenesis and up-regulated obviously in various types of tumor cells and activated endothelial cells. Since the arginine-glycine-aspartic acid (RGD) tripeptide sequence can bind to integrin αvβ3 with high affinity and specificity, RGD PET/CT may be helpful to evaluate the biological and metabolic activity status during angiogenesis. However, 18F-ALF-NOTA-PRGD2 PET/CT as response biomarker for antiangiogenic therapy has not been fully proved and is still without universal understanding according to current publications. Apatinib (YN968D1) is the first orally antiangiogenic drug targeting VEGFR-2 tyrosine kinase.In the current study, investigators propose to evaluate the feasibility of 18F-RGD PET/CT in monitoring efficacy and adverse events of apatinib in malignancies. Patients confirmed malignancies histopathologically will be prospectively enrolled in the study. All patients provided written informed consent prior to enrollment. Patients will receive apatinib therapy, and undergo 18F-RGD PET/CT scans berore and after first cycle of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of malignancies
* Scheduled for second- or third-line apatinib therapy
* Karnofsky performance status (KPS) ≥70
* Measurable primary tumors according to Response Evaluation Criteria in Solid Tumors (RECIST)

Exclusion Criteria:

* Active infection, myocardial infarction within 6 months, symptoms of heart disease, including unstable angina, congestive heart failure or uncontrolled arrhythmias, immunosuppressive therapy
* The claustrophobic patients and patients with implanted metal objects
* The pregnancy
* Inability to complete the required examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2018-01-28 (Actual); Study Completion 2018-01-28 (Actual)

PRIMARY OUTCOMES:
Tumor response defined by RECIST criteria | At 1 month of the study
  Tumor response will be evaluated as complete response or partial response or stable disease or PD according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

SECONDARY OUTCOMES:
Days from the start of therapy to disease progression or death due to any cause | At 6 months of the study
  Progression free survival (evaluated by RECIST criteria), defined as the interval from start of therapy to investigator-assessed progression or death due to any cause, whichever occurs first or lost of follow-up.
Days from the start of therapy to death due to any cause | Up to 12 months
  Overall survival is the time interval from the start of therapy to death due to any reason or lost of follow-up.
Treatment-Related Adverse Events as Assessed by CTCAE | Through study completion, an average of 6 months
  Common Terminology Criteria for Adverse Events （CTCAE）

CONTACTS AND LOCATIONS:
Overall Officials: Shuanghu Yuan, MD;PhD, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No